CLINICAL TRIAL: NCT01097980
Title: The Efficacy of Trazodone for Selective Serotonin Reuptake Inhibitor-induced Sexual Dysfunction
Brief Title: Trazodone for SSRI-sexual Dsyfunction
Acronym: T-SSRI-SD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beitou Armed Forces Hospital, Taipei, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuo-Tung Chiang, Department of Psychiatry, Beitou Armed Forces Hospital, Taipei, Taiwan
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT098-02; CAD-BAFH-M99 (Other Grant/Funding Number: CAD-BAFH-M99)
Record Dates: First submitted 2010-03-28; First posted 2010-04-02 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Sexual Dysfunction
Keywords: trazodone; SSRI; sexual dysfunction; 5-HT2A polymorphism
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trazodone (Experimental): Trazodone versus placebo in a randomized, double-blind manner
  Interventions: Drug: Trazodone
- Placebo (Placebo Comparator): Patients received placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trazodone — 50 mg/d trazodone was upwardly titrated to 100 mg/d over one week and then maintained
  Arms: Trazodone
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the efficacy of trazodone in the treatment of selective serotonin reuptake inhibitor(s) associated sexual dysfunction. The secondary domains assessed were the relationship between 5-HT2A polymorphism and treatment efficacy.

ELIGIBILITY:
Inclusion criteria were:

1. 20-65 years of age,
2. receiving SSRI treatment for more than four weeks,
3. minimal dose of fluoxetine, paroxetine, and citalopram are 20 mg/d, minimal dose of fluvoxamine and sertraline are 50 mg/d, and minimal dose of escitalopram is 10mg/d,
4. developing sexual dysfunction based on the definition of Arizona Sexual Experience-Chinese Version.

Exclusion criteria were:

1. receiving other antidepressant agents,
2. receiving antipsychotics,
3. having a currently unstable medical condition such as unstable angina or uncontrolled diabetes,
4. having any serious medical condition that affects sexual functioning such as epilepsy, serious head injury, brain tumor, HIV infection, Parkinson's disease, dementia, multiple sclerosis, or other neurological disorder,
5. being pregnant or planning to become pregnant during the study period,
6. experiencing psychotic symptoms,
7. being comorbidity with substance abuse, (8) developing sexual dysfunction before receiving SSRIs treatment.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The differences between trazodone and placebo in the Arizona Sexual Experiences Scale-Chinese Version scale at the end of week 6 were used as the primary study outcomes. | week 0 and week 6

SECONDARY OUTCOMES:
The association between 5-HT2A polymorphism and the changes in Arizona Sexual Experiences Scale-Chinese Version scale were evaluated. | week 6
  The secondary domains assessed were the difference between trazodone and placebo in the Clinical Global Impression scale, 10-point Visual Analogue Scale, Hamilton Depression Rating Scale, and Hamilton Anxiety Rating Scale at the end of week 6. Besides, relationships between 5-HT2A polymorphism and the changes in Arizona Sexual Experiences Scale-Chinese Version scale were also evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Tung Chiang, M.D., Study Director — Department of Psychiatry, Beitou Armed Forces Hospital, Taipei, Taiwan
Locations (1):
- Department of Psychiatry, Beitou Armed Forces Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Stryjer R, Spivak B, Strous RD, Shiloh R, Harary E, Polak L, Birgen M, Kotler M, Weizman A. Trazodone for the treatment of sexual dysfunction induced by serotonin reuptake inhibitors: a preliminary open-label study. Clin Neuropharmacol. 2009 Mar-Apr;32(2):82-4. doi: 10.1097/WNF.0B013E31816D1CDC. PMID 18978492